CLINICAL TRIAL: NCT03606798
Title: Multidisciplinary and Personalized Care of Behavioral Disorders in Frontotemporal Lobar Degeneration.
Acronym: DLFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX2015/06
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Frontotemporal Lobar Degeneration
Keywords: Frontotemporal Lobar Degeneration; Behavioral disorders
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary and personalized care (Experimental): Personalized care and proposals bring by a team of experts : neurologists ; geriatrician ; psychologist.
  Interventions: Other: 3 Home visits made by a psychologist
- Reference care (No Intervention): Standard clinical evaluations of patient with Frontotemporal Lobar Degeneration.

INTERVENTIONS:
Other: 3 Home visits made by a psychologist — Patient and caregiver interviews with a psychologist at home
  Arms: Multidisciplinary and personalized care

SUMMARY:
Fronto-Temporal Lobar Degeneration (FTLD) refers to 3 categories of neurodegenerative diseases generally occurring between 55 and 65 years: Fronto-Temporal Dementia(FTD), Primary Progressive Aphasia (PPA), Semantic Dementia (SD). Clinical expression is substantially variable among individuals, but in most cases, behavioural disorders and personality changes are prominent. FTLD is poorly known by general public including health care professionals. Currently, the French health system does not meet the needs and expectations of patients and their families

DETAILED DESCRIPTION:
Patients with FTLD and their caregivers need to be recognized and supported through specific and tailored made actions provided by expert teams. The main objective of our study is to evaluate the effectiveness of a 6-month personalized multidisciplinary care provided to the dyad FTLD patient and caregiver on patient's behavioural disorders. The secondary objectives are to assess the impact of this program on patient's cognitive deterioration, functional autonomy and behavioral problems, as well as caregiver's depressive symptomatology and sense of competence

ELIGIBILITY:
Inclusion criteria:

Patients

* Fronto-Temporal Lobar Degeneration diagnoses
* Men or women aged 18 and over

Caregiver

• Spouse, brother, sister, child living at patient's home and can provide the medical team of reliable information on the status of their parent.

Exclusion criteria :

Patient

* Patient institutionalized
* Pregnant or breast-feeding woman
* Psychotic syndrome
* Severe and unstable general medical condition
* Patient bedridden

Caregiver

* Persons under legal protection
* Severe and unstable general medical condition
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | 6 months
  Assessment of neuropsychiatric symptomatology

SECONDARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | 12 months
  Assessment of neuropsychiatric symptomatology
Mini Mental State Examination | 6 months and 12 months
Frontal Behavioral Inventory | 6 months and 12 months
Frontal Assessment Battery | 6 months and 12 months
Geriatric Depression Scale Score ( From 0 to 30) | 6 months and 12 months
  Score : 0 - 5 : normal Score : 5 - 9 : light depression Score : 10 - 30 : severe depression
Sense of Competence Questionnaire (SCQ) | 6 months and 12 months
Quality of Life Questionnaire (QoL-AD) | 6 months and 12 months
Hierarchical scale of internality for elderly people (EHIPA) score ( From 0 to 22) | 6 months and 12 months
  The score varies from 0 to 22. A high score corresponding to an important internality

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François DARTIGUES, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No